CLINICAL TRIAL: NCT07003256
Title: An Observational Study on the Promotion of Platelet Recovery by Romiplostim During Haploidentical Hematopoietic Stem Cell Transplantation
Brief Title: Observational Study: Romiplostim for Platelet Recovery in Haploidentical HSCT
Status: Enrolling by invitation | Type: Observational
Sponsor: Haikou Affiliated Hospital of Central South University Xiangya School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: JVKY2024-0101015002
Record Dates: First submitted 2025-05-15; First posted 2025-06-04 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Thalassemia in Children
Keywords: Thalassemia; Romiplostim; HSCT
MeSH Terms: conditions — Thalassemia | interventions — romiplostim

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- experimental group: After transplantation + 6 days, the subcutaneous injection of roprastine 3ug/kg was started, and the number of platelets in the machine-taken platelet suspension was increased by 2 µg/kg per week, and the maximum dose was 10 μg/kg. Discontinued until platelets rose to 100 × 109/L. If platelets ≤ 20 X 109/L were used for + 20 days, roprastine combined with atropopa 25mg was given orally once a day. Patients were given 1 therapeutic dose of fresh machine-taken platelet suspension when platelets were ≤ 20 X 109/L, or when there was active bleeding at 21~ 50 × 109/L. The number of platelets in the machine-taken platelet suspension per therapeutic dose was > 2.5 × 1011. If not implanted at + 28 days after transplantation, re-transplantation is required, and roprastine is considered ineffective.
  Interventions: Drug: Romiplostim

INTERVENTIONS:
Drug: Romiplostim — After transplantation + 6 days, the subcutaneous injection of roprastine 3ug/kg was started, and the number of platelets in the machine-taken platelet suspension was increased by 2 µg/kg per week, and the maximum dose was 10 μg/kg. Discontinued until platelets rose to 100 × 109/L. If platelets ≤ 20 X 109/L were used for + 20 days, roprastine combined with atropopa 25mg was given orally once a day. Patients were given 1 therapeutic dose of fresh machine-taken platelet suspension when platelets were ≤ 20 X 109/L, or when there was active bleeding at 21~ 50 × 109/L. The number of platelets in the machine-taken platelet suspension per therapeutic dose was > 2.5 × 1011. If not implanted at + 28 days after transplantation, re-transplantation is required, and roprastine is considered ineffective.
  Other Names: Nplate

SUMMARY:
The objective of this observational study is to explore the long-term effects of roprastine given to promote platelet implantation in hematopoietic stem cell hemicongruent transplantation in children with thalassemia. The main questions it aimed to answer is:

Is roprastine safe and effective for platelet implantation in children with thalassemia hemicongruent transplantation? Participants who have already received roprastine as part of routine medical care for hematopoietic stem cell hemicongruent transplantation in children with thalassemia will answer online survey questions about the effects of their platelet implantation within 8 weeks.

DETAILED DESCRIPTION:
Allogeneic hematopoietic stem cell transplantation is an important, if not the only, means of curing many diseases of the blood system. Thrombocytopenia after transplantation seriously affects the long-term survival rate of patients. allo - The incidence of thrombocytopenia in HSCT patients is 5-20% (< 20 x 10 ^ 9/L), increasing the risk and cost of treatment. There are currently few studies on the promotion of platelet growth in children with thalassemia. Repeated infusion of platelet suspension can lead to many adverse consequences, including blood transfusion reactions, platelet homeoimmune responses, and transfusion-associated virus infections. There is a black box warning of liver toxicity in eltropopa, and the incidence of real-world liver toxicity is 11.8%. Transplant patients are prone to diarrhea, which affects the absorption of oral platelet-raising drugs. Daily subcutaneous injection increases children's pain and poor tolerance. However, the long-acting platelet-raising drugs once after transplantation are well tolerated in children with thalassemia transplantation, and the efficacy is worth looking forward to. Up to now, there is a lack of relevant clinical data on the application of roprastine to promote platelet recovery in children with thalassemia hemiphase transplantation. Therefore, this study aimed to explore the observational study of roprastine to promote platelet implantation in children with thalassemia hemiphase transplantation, and to explore the efficacy and safety of the drug.

ELIGIBILITY:
Inclusion Criteria:

* After undergoing Mediterranean gene testing, reviewing the history of blood transfusions, and conducting a blood routine examination, the patient was diagnosed with severe thalassemia.
* Children aged 2 - 17 years old.
* Agree to the haploidentical transplantation, and the team has evaluated that there are no transplantation contraindications.

Exclusion Criteria:

* There is a fully matched donor, and transplantation with a half - matched donor is not agreed.
* For donors and recipients, the transaminase is more than twice the normal value.
* Donor specific antibody Greater than 5000, and after antibody treatment, it should not be lower than 3000.
* Positive for hepatitis B DNA.
* There is an active infection.
* After evaluation by the transplantation team, there are contraindications for transplantation.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged 2 - 17 years old who were diagnosed with severe thalassemia at Haikou People's Hospital and received haploidentical hematopoietic stem cell transplantation.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Platelet recovery time | From enrollment to 28 days after transplantation
  The time at nodes such as platelet >20×10^9/L, 50×10^9/L and 100×10^9/L
Platelet transfusion volume | From enrollment to 28 days after transplantation
  The required dosage of platelet suspension

SECONDARY OUTCOMES:
Adverse drug reaction rate | From enrollment to 28 days after transplantation
  The rate of adverse drug reactions occurring during the follow-up period
Bleeding incidence rate | From enrollment to 28 days after transplantation
  The incidence rate of bleeding that occurred during the follow-up period
Thrombosis incidence rate | From enrollment to 28 days after transplantation
  The incidence rate of thrombosis occurring during the follow-up period
Survival rate | From enrollment to 28 days after transplantation
  The survival rate of patients after transplantation medication
Recurrence - free survival rate | From enrollment to 28 days after transplantation
  The survival rate of patients without recurrence of the disease after using the drug
Transplant - related mortality | From enrollment to 28 days after transplantation
Major transplant-related complications | From enrollment to 28 days after transplantation
Cause of death | From enrollment to 28 days after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoyang Yang, MD, Principal Investigator — Department of Hematology, Haikou People's Hospital
Locations (1):
- Haikou Affiliated Hospital of Central South University Xiangya School of Medicine, Haikou, Hainan, China

IPD SHARING:
Plan to Share IPD: No
The IPD encompasses highly sensitive and confidential data that was collected through significant investment of our resources, both in terms of time and funding. This data is integral to our ongoing research initiatives, which are at a crucial stage of development. Premature sharing could disrupt our research timelines and strategic plans. Additionally, we have not yet established comprehensive safeguards to ensure that the data will be used appropriately by external researchers. Without proper protocols in place, there is a risk of misuse or misinterpretation of the data, which could lead to inaccurate research outcomes and potential reputational damage to our institution. For these reasons, we have decided not to share the IPD at this time.